CLINICAL TRIAL: NCT03191266
Title: Transcranial Magnetic Stimulation for the Treatment of Veterans With Alcohol Use Disorders
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D2303-R; 1I01RX002303-01A2 (NIH)
Record Dates: First submitted 2017-06-02; First posted 2017-06-19 (Actual); Results first posted 2026-01-28 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Alcohol Use Disorder
Keywords: repetitive transcranial magnetic stimulation; alcohol use disorder; neuroimaging; relapse; Veterans
MeSH Terms: conditions — Alcoholism; Recurrence

STUDY DESIGN:
Intervention Model Description: A double-blind randomized clinical trial with two groups: Active rTMS Treatment Group (Active rTMS) - will receive four to five treatments (two treatments per day) each week for 2 weeks. Sham Control Treatment group (i.e., identical rTMS experimental procedure, but no active stimulation) will receive the same frequency and duration of rTMS sessions. The proposed rTMS protocol is consistent with the FDA approved treatment regimen employed for major depressive disorders.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: A double-blind randomized clinical trial with two groups: Active rTMS Treatment Group (Active rTMS) - will receive four to five treatments (two treatments per day) each week for 2 weeks. Sham Control Treatment group (i.e., identical rTMS experimental procedure, but no active stimulation) will receive the same frequency and duration of rTMS sessions.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- active rTMS (Active Comparator): Active rTMS will receive an intermittent rTMS stimulation protocol.
  Interventions: Device: Active rTMS
- sham rTMS (Sham Comparator): Sham rTMS will receive all conditions except the actual intermittent theta burst rTMS stimulation.
  Interventions: Device: Sham rTMS

INTERVENTIONS:
Device: Active rTMS — Active rTMS will receive an intermittent rTMS stimulation protocol.
  Arms: active rTMS
Device: Sham rTMS — Sham rTMS will receive all conditions except the actual intermittent theta burst rTMS stimulation.
  Arms: sham rTMS

SUMMARY:
At least 60% of Veterans with an alcohol use disorder will relapse within 6 months of treatment, irrespective of the type of treatment they receive. This indicates that currently available interventions for treating AUD in Veterans are not effective in helping them achieve long-term sobriety. Repetitive transcranial magnetic stimulation (rTMS) is a brain stimulation method that is at the forefront of innovative, non-invasive, and safe treatments for AUD. However, there have been no studies that specifically determined the effectiveness of rTMS treatment for Veterans with AUD. This project will evaluate the effectiveness of rTMS treatment in promoting long-term abstinence in Veterans suffering from AUD. Assisting Veterans in achieving long-term and sustained sobriety is critical because it is associated with the best medical, cognitive, psychiatric, and psychosocial recovery from AUD.

DETAILED DESCRIPTION:
Due to COVID-19 restrictions, active recruiting was suspended 31MAR20. Recruitment resumed 1SEP21

The purpose of this study is to evaluate the efficacy of intermittent theta burst repetitive transcranial magnetic stimulation (rTMS) as a treatment for Veterans with an alcohol use disorder (AUD) to decrease the exceedingly high rate of relapse associated with this condition.

At least 60% of those with AUD will experience a major relapse period within 6 months of treatment, irrespective of the intervention (psychosocial and/or pharmacological) employed. Consequently, the high prevalence of AUD and relapse following treatment in Veterans is associated with substantial resource allocation and costs for the DVA Health Care System. Current pharmacological and psychosocial interventions demonstrate only a moderate level of efficacy, which is reflected in the high rate of relapse in AUD.

rTMS is a neurostimulation method that is at the forefront of innovative, non-invasive, and safe treatments for AUD, and the disorders that commonly co-occur with AUD. To reduce the high rate of relapse in Veterans with AUD, it is necessary for interventions to more effectively address the associated neurobiological dysfunction and salient co-occurring conditions. Accordingly, additional rigorously controlled studies are required to determine if intermittent theta burst rTMS is an effective treatment for Veterans with AUD.

Participants will be recruited from VA Palo Alto Health Care System (VAPAHCS) residential substance abuse treatment clinics A double-blind randomized clinical trial with two groups: Active rTMS Treatment Group (Active rTMS) - will receive five treatments (two treatments per day) per week for 2 weeks. Sham Control Treatment group (i.e., identical rTMS experimental procedure, but no active stimulation) will receive the same frequency and duration of rTMS sessions. The proposed rTMS protocol is consistent with the FDA approved treatment regimen employed for major depressive disorders at the VAPAHCS MIRECC. Magnetic resonance imaging (MR) will be completed pre and post rTMS treatment and used to localize the left DLPFC in each participant to optimize rTMS for this region. Active and Sham rTMS groups will complete predictive measures [i.e., MR measures of anterior frontal glutamate level, blood flow, and tissue volume, diffusion tensor imaging, functional connectivity, task-based fMRI] and other outcome measures (i.e., measures of craving, mood, anxiety, neurocognition) immediately pre- and post-completion of the 2 weeks of rTMS sessions. Genetic markers (i.e., brain derived neurotrophic factor plasma levels and polymorphisms) will also be collected. Neuroimaging and genetic measures are necessary to establish potential biomarkers for prediction of rTMS treatment response, which is requisite for therapeutic optimization. For the 6 months following completion of active or sham rTMS treatment, participants will be contacted monthly, via telephone or in person, to complete a brief standardized measure of alcohol and substance use, craving, and psychiatric symptomatology to assess for changes in these variables over the previous 30 days.

This project will deliver completely novel data on the efficacy of intermittent theta burst rTMS for Veterans with AUD during the first 6 months following treatment. Monitoring over the entire first 6 months following treatment is crucial, given relapse within the first 6 months of treatment is robustly related to poor psychosocial functioning over the ensuing 1-3 years. The ultimate goal of this proposal is provide treatment that more effectively promotes sustained abstinence in the Veteran with AUD, as extended abstinence is robustly associated with optimum biomedical, neuropsychological, psychiatric, and psychosocial recovery and functioning.

ELIGIBILITY:
Inclusion Criteria:

* The study will be open to male and females, regardless of race and ethnic origin, who are in active treatment for an alcohol use disorder (AUD).
* Meet Diagnostic and Statistical Manual of Mental Disorders, 5th Edition criteria for AUD, and alcohol is self-identified as primary substance of misuse.
* Actively in treatment at VA Palo Alto HCS Addiction Treatment Service, and able to read, verbalize understanding, and voluntarily sign the Informed Consent Form prior to participation in study procedures.
* Participants will be accepted if taking medications specifically for the treatment of MDD, cigarette smoking, or for other psychiatric conditions.

  * as long as the medications are not documented to lower seizure threshold
  * must be stable on any psychotropic medication for at least 1 month prior to enrollment
  * it would be clinically contraindicated to require participants to discontinue such medications for research.
* Participants will be abstinent from alcohol and non-prescribed substances for at least 7 consecutive days prior to active or sham rTMS and no participant demonstrates active acute withdrawal symptoms.

Exclusion Criteria:

Psychiatric:

* History of Schizophrenia Spectrum Disorders
* Bipolar Disorders
* A current substance use disorder that exceeds the severity of the AUD

  * based on DSM-5 diagnostic criteria
* Current use of an FDA approved medication for treatment of AUD, i.e.:

  * disulfiram
  * acamprosate
  * naltrexone
* Active current suicidal intent or plan

  * patients with a previous clinical flag for risk for suicide will be required to have an established safety plan involving their primary psychiatrist and the treatment team before entering the clinical trial
* Any form of previous rTMS or electroconvulsive treatment

Biomedical:

* Including but not limited to uncontrolled thyroid disease
* Unstable congestive heart failure
* Angina
* Other severe cardiac illness as defined by treatment regimen changes in the prior 3 months
* Cerebrovascular accident
* Cancer if < 1 year since end of treatment
* Unstable diabetes
* COPD requiring oxygen supplementation
* Alzheimer's disease
* Parkinson's disease
* Any biomedical implants with ferromagnetic content
* Neurostimulation devices
* Cardiac pacemakers or any magnetic resonance contraindications
* Traumatic brain injury with self-reported or observed loss of consciousness > 30 minutes
* Any primary or traumatically induced seizure disorder

General:

* Lack of fluency in English
* Wechsler Adult Reading Test below the 7th percentile, i.e.:

  * moderate or greater impairment in estimated general intelligence
* Females who are pregnant or actively attempting pregnancy

  * conservative exclusion for magnetic resonance research
* Current use of any medication or substance that is documented to lower seizure threshold or has been identified as a contraindication for rTMS treatment

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2018-04-15 (Actual); Primary Completion 2024-06-28 (Actual); Study Completion 2024-06-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Timothy C. Durazzo, PhD, Principal Investigator — VA Palo Alto Health Care System, Palo Alto, CA
Locations (1):
- VA Palo Alto Health Care System, Palo Alto, CA, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Final datasets in machine-readable format will be submitted to PubMed Central, which will permit the easiest access All participants will be assigned a subject code, which will have no relationship to any aspect of identifiable private information. Therefore, the data associated with each participant will be completely de-identified. There will be no mechanism by which public users will be able to re-identify participant data (e.g., name, address) with the subject code.

REFERENCES:
- [Derived] Durazzo TC, McNerney MW, Hansen AM, Gu M, Sacchet MD, Padula CB. BDNF rs6265 Met carriers with alcohol use disorder show greater age-related decline of N-acetylaspartate in left dorsolateral prefrontal cortex. Drug Alcohol Depend. 2023 Jul 1;248:109901. doi: 10.1016/j.drugalcdep.2023.109901. Epub 2023 Apr 28. PMID 37146499

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Eighty-eight Veterans with alcohol use disorder, from a residential treatment program at the VA Palo Alto Health Care System, completed an in-person screen for study eligibility.Thirty-four individuals were not eligible for participation; the most common reasons for exclusion were a history of bipolar or schizophrenia spectrum disorders or moderate or greater severity traumatic brain injury. Five other participants were eligible, but declined to complete the 2-week study procedure.
Pre-assignment Details: Eighty-eight Veterans with alcohol use disorder, completed an in-person screen for study eligibility. Thirty-four individuals were not eligible for participation. Five other participants were eligible, but three declined, not wishing to complete neuroimaging procedures, and two did not wish to complete the approximately 2-week iTBS procedure. The final participant group consisted of 49 individuals.
Period: Overall Study
Arm/Group | Active rTMS | Sham rTMS
Started | 25 | 24
Completed | 22 | 22
Not Completed | 3 | 2
Not completed — Space occupying lesion on MRI; PI removed participant after randomization, but before TMS initiation | 0 | 1
Not completed — Withdrawal by Subject | 3 | 1

BASELINE CHARACTERISTICS:
Population: Reported numbers include all participants randomized to active or sham rTMS.
Groups:
- Total: Total of all reporting groups
Arm/Group | Active rTMS | Sham rTMS | Total
Number analyzed (Participants) | 25 | 24 | 49
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.6 (13.8) | 51.3 (13.8) | 51.0 (13.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 1
  Male | 25 | 23 | 48
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Latino/Hispanic
  Participants
    Hispanic or Latino | 6 | 5 | 11
    Not Hispanic or Latino | 19 | 19 | 38
    Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3 | 0 | 3
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 3 | 5 | 8
  White | 18 | 17 | 35
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Formal education [Mean (Standard Deviation); unit: years] — Years of formal education
  years | 14.3 (2.4) | 14.0 (1.6) | 14.2 (2.0)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Abstained From Alcohol
Description: For the 6 months following completion of active or sham rTMS treatment, participants were contacted monthly, via telephone or in person, to complete a brief standardized measure of alcohol and substance use, and psychiatric symptoms to assess for changes in these variables over the previous 30 days.
Time Frame: 6 months following last TMS session
Measure: Count of Participants; unit: Participants
Arm/Group | Active rTMS | Sham rTMS
Number analyzed (Participants) | 22 | 22
Participants | 13 | 9
Statistical Analysis 1: Comparison: Active rTMS vs Sham rTMS; Test type: Other; p = 0.05, Regression, Logistic — Logistic regression tested the hypothesis that the odds of continuous abstinence was greater, at 6 months following post-assessment, in the Active (n = 22) versus the Sham (n = 22) group. P < 0.05 considered statistically significant; Covariate included average drinks per day 3-months prior to study; Odds Ratio (OR) = 4.4, 95% CI 2-sided [1.0 to 18.9]

2. Secondary Outcome: Glutamate Concentration in the Left Dorsolateral Prefrontal Cortex (as Measured With Single Voxel Spectroscopy)
Description: Determine if baseline glutamate level can serve as a biomarker to differential those participant, in the active rTMS group who main continuous abstinence versus those who resumed alcohol consumption.
Time Frame: Baseline
Population: This grouping within the active rTMS arm (Abstinent or Resumed alcohol consumption during the 6 month follow-up period) was conducted to determine if baseline glutamate level can serve as a biomarker to differential those participants, in the active rTMS group who main continuous abstinence versus those who resumed alcohol consumption. The investigators did not hypothesize that baseline glutamate would predict outcome (abstinent vs. resumed) in the sham rTMS group.
Measure: Mean (Standard Deviation); unit: mmol/L
Groups:
- Active rTMS (Abstinent): Group represents glutamate level (scaled to water, adjusted for cerebrospinal fluid concentration, institutional units) in the left dorsolateral prefrontal cortex, at baseline, in active participants who maintained continuous abstinence (Abstained, n = 8) over the 6-month follow-up interval. Due to MR scanner downtime due to upgrades and the COVID-19 pandemic, only 14 of 22 active participants completed single volume spectroscopy.
- Active rTMS (Resumed): Group represents glutamate level (scaled to water, adjusted for cerebrospinal fluid concentration, institutional units) in the left dorsolateral prefrontal cortex, at baseline, in active participants who resumed alcohol consumption (Resumed, n = 6) during the 6-month follow-up interval. Due to MR scanner downtime due to upgrades and the COVID-19 pandemic, only 14 active participants completed single volume spectroscopy.
Arm/Group | Active rTMS (Abstinent) | Active rTMS (Resumed)
Number analyzed (Participants) | 8 | 6
mmol/L | 26.2 (2.6) | 19.7 (3.0)
Statistical Analysis 1: Comparison: Active rTMS (Abstinent) vs Active rTMS (Resumed); Comparison of baseline left dorsolateral prefrontal cortex (DLPFC) glutamate level in participants in the active rTMS group that maintained continuous abstinence over 6 months (Abstinent) versus those who resumed alcohol consumption (Resumed). Higher glutamate level is considered neurobiologically advantageous; Test type: Other; p = 0.11, generalized linear model — p < 0.05 considered statistically significant; Mean Difference (Final Values) = 6.4, 95% CI 2-sided [-1.4 to 14.3], Standard Error of Mean 4.01

3. Secondary Outcome: Volume in Anterior Frontal Cortical Regions (as Measured With FreeSurfer)
Description: Determine if volume in anterior frontal cortical regions can serve as biomarkers to predict rTMS treatment response in Veterans with AUD who receive active TMS. Specific regions of interest were the left caudal and rostral middle frontal gyrus and left superior frontal gyrus because these regions correspond to the rTMS anatomical target.
Time Frame: Baseline
Population: This grouping within the active rTMS arm (Abstinent or Resumed alcohol consumption during the 6 month follow-up period) was conducted to determine if baseline left caudal and rostral middle frontal and left superior frontal gyri could gyrus serve as a biomarker to differential those participants, in the active rTMS group, who main continuous abstinence versus those who resumed consumption. We did not hypothesize baseline volumes would predict outcome (abstinent vs. resumed) in the sham group.
Measure: Mean (Standard Deviation); unit: Volume in cubic millimeters
Groups:
- Active rTMS (Abstinent): Group represents volumes in cubic millimeters (adjusted for age and total intracranial volume) in the left caudal and rostral middle frontal gyrus and left superior frontal gyrus, in active participants, who maintained continuous abstinence (Abstained, n = 9), over the 6-month follow-up interval. Due to MR scanner downtime due to upgrades and the COVID-19 pandemic, only 17 of 22 active participants completed structural magnetic resonance imaging.
- Active rTMS (Resumed): Group represents volumes in cubic millimeters (adjusted for age and total intracranial volume) in the left caudal and rostral middle frontal gyrus and left superior frontal gyrus, in active participants, who resumed alcohol consumption (Resumed, n = 8), during the 6-month follow-up interval. Due to MR scanner downtime due to upgrades and the COVID-19 pandemic, only 17 active participants completed structural magnetic resonance imaging.
Arm/Group | Active rTMS (Abstinent) | Active rTMS (Resumed)
Number analyzed (Participants) | 9 | 8
Volume in cubic millimeters
  left caudal middle frontal gyrus | 6587 (1029) | 6236 (933)
  left rostral middle gyrus frontal gyrus | 14778 (1963) | 14071 (2549)
  left superior frontal gyrus | 23503 (2693) | 21086 (2729)
Statistical Analysis 1: Comparison: Active rTMS (Abstinent) vs Active rTMS (Resumed); Comparison of baseline left caudal middle frontal gyrus volume (cubic millimeters) in participants in the active rTMS group that maintained continuous abstinence over 6 months (Abstinent) versus those who resumed alcohol consumption (Resumed). Larger volumes are considered neurobiologically advantageous; Test type: Other; p = 0.92, generalized linear model — P < 0.05 considered statistically significant; covariates included age and total intracranial volume; Mean Difference (Final Values) = 58, 95% CI 2-sided [-1258 to 1142], Standard Error of Mean 556
Statistical Analysis 2: Comparison: Active rTMS (Abstinent) vs Active rTMS (Resumed); Comparison of baseline left rostral middle frontal gyrus volume (cubic millimeters) in participants in the active rTMS group that maintained continuous abstinence over 6 months (Abstinent) versus those who resumed alcohol consumption (Resumed). Larger volumes are considered neurobiologically advantageous; Test type: Other — age and intracranial volume were covariates; p = 0.56, generalized linear model — P < 0.05 considered statistically significant; Mean Difference (Final Values) = 518, 95% CI 2-sided [-1361 to 2399], Standard Error of Mean 870
Statistical Analysis 3: Comparison: Active rTMS (Abstinent) vs Active rTMS (Resumed); Comparison of baseline left superior frontal gyrus volume (cubic millimeters) in participants in the active rTMS group that maintained continuous abstinence over 6 months (Abstinent) versus those who resumed alcohol consumption (Resumed). Larger volumes are considered neurobiologically advantageous; Test type: Other; p = 0.49, generalized linear model — age and intracranial volume were covariates; Mean Difference (Final Values) = 942, 95% CI 2-sided [-3549 to 1663], Standard Error of Mean 1206

4. Secondary Outcome: BDNF Polymorphisms (as Measured With TaqMan Genotyping Assays or Similar Assays)
Description: Determine if BDNF polymorphisms (rs6265) can serve as biomarkers to predict rTMS treatment response in Veterans with AUD. Analysis focused on comparing Val homozygote frequency, in active rTMS arm participants, who maintained continuous abstinence (Abstinent) versus those who resumed alcohol consumption (Resumed) over the 6-month follow-up period. There were a limited number of participants who completed the genotyping procedure; therefore, results are likely not generalizable.
Time Frame: Baseline
Population: Analysis was conducted to determine if BDNF polymorphisms (rs6265) can serve as biomarkers to predict rTMS treatment response in Veterans with AUD. Analysis focused on comparing Val homozygote frequency, in active rTMS arm participants, who maintained continuous abstinence (Abstinent) versus those who resumed alcohol consumption (Resumed) over the 6-month follow-up period. We did not have specific hypotheses about BDNF polymorphism rs6265 for abstinence or resumption of alcohol in sham arm.
Measure: Count of Participants; unit: Participants
Groups:
- Active rTMS (Abstinent): Group represents frequency of BDNF rs6265 Val/Val homozygotes in active participants who maintained continuous abstinence (Abstained, n = 7) over the 6-month follow-up interval.
- Active rTMS (Resumed): Group represents frequency of BDNF rs6265 Val/Val homozygotes in active participants who maintained continuous abstinence, in active participants who resumed alcohol consumption (Resumed, n = 4) during the 6-month follow-up interval.
Arm/Group | Active rTMS (Abstinent) | Active rTMS (Resumed)
Number analyzed (Participants) | 7 | 4
Participants | 5 | 4
Statistical Analysis 1: Comparison: Active rTMS (Abstinent) vs Active rTMS (Resumed); Test type: Other; p = 0.24, Chi-squared, Corrected — P < 0.05 considered statistically significant; Asymptotic Significance (2-sided) = 1.4

ADVERSE EVENTS:
Time Frame: 1 year post study completion for each participant.
Description: Participant was the under the care of VA clinicians at the time of death and was formally screened for suicidal ideation/intent by different VA clinicians on 9 and 3 days prior to death and denied any suicidal ideation.
Arm/Group | Active rTMS | Sham rTMS
All-Cause Mortality (participants affected / at risk) | 0/22 | 1/22
Serious Adverse Events (participants affected / at risk) | 0/22 | 1/22
Other Adverse Events (participants affected / at risk) | 0/22 | 0/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Active rTMS (N=22) | Sham rTMS (N=22)
suicide (Psychiatric disorders) | 0 (0) | 1 (1) — PI was notified that the participant committed suicide 66 days after final rTMS session. Participant was intoxicated at the time of their death. VA/Stanford IRB concluded participant death was unrelated to study interventions.

LIMITATIONS AND CAVEATS:
Due to the extended halt of human subject recruitment during the COVID-19 pandemic, and the Principal Investigator's (TCD) 1.5 year active duty military deployment during the study recruitment phase, the sample size was lower than the 100 used to power the current study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2025-06-27): https://cdn.clinicaltrials.gov/large-docs/66/NCT03191266/Prot_SAP_000.pdf
  • Informed Consent Form (2023-07-27): https://cdn.clinicaltrials.gov/large-docs/66/NCT03191266/ICF_001.pdf